CLINICAL TRIAL: NCT06006260
Title: Changes of Low Anterior Resection Syndrome, Balance Ability, and Quality of Life in Patients with Newly Diagnosed Rectal Cancer.
Brief Title: Changes of Low Anterior Resection Syndrome and Balance Ability in Patients with Rectal Cancer.
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20220197B0
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purposes of this study are to explore the trajectory of symptom distress and balance ability in patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed rectal cancer
2. Patients already know their condition.
3. Aged 20 years and older.
4. Consciously communicate in Mandarin or Taiwanese.
5. Agreed with the interview and had signed the permit.

Exclusion Criteria:

1. Recurrent rectal cancer.
2. KPS of patients less than 80

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients during therapy.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-report Questionnaire | Change from baseline symptom at 2 months
  Show the specific trajectory of LAR Syndrome, psychological distress, fecal incontinence-related QoL, and balance ability based on different tumor locations in patients with rectal cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Gung University, Taoyuan, Kwei-Shan Dist., Taiwan